CLINICAL TRIAL: NCT04273230
Title: Early Detection of Kidney Affection in Non Alcaholic Fatty Liver Diseases(NAFLD)
Brief Title: Kidney Affection in Non Alcaholic Fatty Liver Diseases
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Emad Atta Saad Girgis, Doctor, Assiut University
Other Study IDs: Kidney affection in NAFLD
Record Dates: First submitted 2020-02-14; First posted 2020-02-18 (Actual); Last update posted 2022-02-23 (Actual); Status verified 2020-02

CONDITIONS: Renal Impairment
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Microalbuminuria detection — Detection of microalbumin in urine

SUMMARY:
Early detection of renal affection in patients with non alcaholic fatty liver diseases using microalbuminuria.

DETAILED DESCRIPTION:
With the increasing prevalence of obesity, diabetes mellitus and the metabolic syndrome in the general population, non-alcoholic fatty liver disease (NAFLD) has become the most common cause of chronic liver disease. NAFLD refers to a wide spectrum of liver damage, ranging from simple steatosis to non-alcoholic steatohepatitis, advanced fibrosis and cirrhosis as well hepatocellular carcinoma.

Several large cross-sectional population and hospital-based studies involving both diabetic patients and patients without diabetes have consistently shown that the prevalence of CKD is increased in people with NAFLD . NAFLD and CKD share some common features, including visceral obesity,T2DM, hypertension and metabolic syndrome . The possible link between NAFLD and CKD has recently attracted considerable scientific interest. Establishing a link between liver and kidney injury would enhance the earlier identification of kidney disease and allow for the selection of treatments targeting both liver and kidney disease with potentially relevant preventive and therapeutic implications . The ultimate goal of identifying patients with established but also with early kidney damage is to prevent disease progression and minimize complications, to promote quality of life and improve survival .

Many recent studies, including the meta-analysis from Musso et al. suggest that individuals with NAFLD should be screened for CKD by estimation of GFR and urinalysis even in the absence of classical risk factors for CKD, particularly if NASH and/or advanced fibrosis are suspected . Early recognition of impaired kidney function in patients with NAFLD, may also allow drug dosage adjustment, thus preventing drug accumulation especially in those being treated for obesity associated co-morbidities.

Chronic kidney disease (CKD) is defined by the presence of reduced glomerular filtration rate (GFR <60 mL/min/1.73 m2)and/or evidence of kidney damage (usually indicated by albuminuria or proteinuria) for 3 or more months . On the other hand kidney failure is defined as a GFR of less than 15 mL/min per 1.73 m2,or the need for treatment with dialysis or transplantation . In clinical practice the most common tests for CKD diagnosis include eGFR estimated from the serum creatinine concentration and albuminuria from the urinary albumin-to-creatinine ratio (ACR). The importance of eGFR and albuminuria as diagnostic tools becomes obvious by their use in classification of CKD patients in stages .On the basis of GFR the disease is classified into five stages:more than 90 mL/min per 1.73 m2(stage 1), 60-89 mL/min per1.73 m2(stage 2), 30-59 mL/min per 1.73 m2(stage 3), more specific 45-59 mL/min per 1.73 m2(stage 3a) and 30-44 mL/min per1.73 m2(stage 3b), 15-29 mL/min per 1.73 m2(stage 4) and less than 15 mL/min per 1.73 m2(stage 5) .

Albuminuria as a marker of kidney damage is characterized by increased glomerular permeability and urine ACR > 30 mg/g. The normal urinary ACR in young adults is <10 mg/g. Urine ACR categories 10-29, 30-300and >300 mg are high normal, high, and very high, respectively.Urine ACR >2000 mg/g is accompanied by signs and symptoms of nephrotic syndrome (low serum albumin, edema, and high serum cholesterol)

ELIGIBILITY:
Inclusion Criteria:

* All patients with fatty liver disease diagnosed by abdominal ultrasonogarphy .
* All patients with fatty liver disease diagnosed by lab investigations.

Exclusion Criteria:

* Diabetic patients
* Hypertensive patients
* patients with chronic kidney disesase
* patient with systemic diseases or chronic liver diseases affecting kidneys.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All pateints with fatty liver diseases diagnosed by ultrasonography and lab investigation
Sampling Method: Non-Probability Sample
Enrollment: 114 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Early detection of kidney affection in non alcaholic fatty liver diseases | Baseline
  Finding patients with non alcaholic fatty liver diseases who develop renal impairment

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Assiut university, Asyut
  - AssiutU, Asyut

REFERENCES:
- [Background] Arase Y, Suzuki F, Kobayashi M, Suzuki Y, Kawamura Y, Matsumoto N, Akuta N, Kobayashi M, Sezaki H, Saito S, Hosaka T, Ikeda K, Kumada H, Ohmoto Y, Amakawa K, Tsuji H, Hsieh SD, Kato K, Tanabe M, Ogawa K, Hara S, Kobayashi T. The development of chronic kidney disease in Japanese patients with non-alcoholic fatty liver disease. Intern Med. 2011;50(10):1081-7. doi: 10.2169/internalmedicine.50.5043. Epub 2011 May 1. PMID 21576832
- [Background] Kiapidou S, Liava C, Kalogirou M, Akriviadis E, Sinakos E. Chronic kidney disease in patients with non-alcoholic fatty liver disease: What the Hepatologist should know? Ann Hepatol. 2020 Mar-Apr;19(2):134-144. doi: 10.1016/j.aohep.2019.07.013. Epub 2019 Sep 23. PMID 31606352
- [Background] Park H, Dawwas GK, Liu X, Nguyen MH. Nonalcoholic fatty liver disease increases risk of incident advanced chronic kidney disease: a propensity-matched cohort study. J Intern Med. 2019 Dec;286(6):711-722. doi: 10.1111/joim.12964. Epub 2019 Aug 23. PMID 31359543